CLINICAL TRIAL: NCT06241157
Title: A Novel Behavior Guidance Technique: "The Pediatric Quiz Game" for the Management of Anxious Children
Brief Title: Pediatric-Quiz Game Behaviour Guidance in Children
Acronym: Pedodontics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: MU_SD_DPD
Record Dates: First submitted 2024-01-05; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Behavior, Child
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: There are two experimental groups. The part containing the first group will be completed first, and then the other group will begin. Same dentist will carry out in the experimental part of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Quiz Game (Experimental): Behavior Guidance Technique (BGT) group (Pedo-Quiz group) Whereas, with the novel BGT so called "The Pediatric-Quiz Game" (PQ), dentists start interacting with children in the waiting room before entering the operating room. It can be defined as "asking children basic questions on colors, animals, fruits and/or cities depending on the age of the child. Each child will be asked to fill out the "Facial Shape Scale" and the "Venham Picture Test" before the procedure. After the session, the Frankl Behavior Scale and the "Patient Evaluation Form" will be filled out by the dentist. Their families (parents/guardians) will be asked to fill out the "Child Fear Assessment Scale-Dental Subscale (CFSS-DSc) before the session. 35 children will be included in the study.Main goal in this sesion is to evaluate in which dental practice step can be progressed in an anxious child by using this new behavior managament technique.
  Interventions: Other: Pediatric Quiz Game
- Control (No Intervention): This group is the control group. Tell-show-do technique, which is a frequently used behavioral management techniques will be used.
  In this group, each child will be asked to fill out the "Facial Shape Scale" and the "Venham Picture Test" before the procedure. After the session, the Frankl Behavior Scale and the "Patient Evaluation Form" will be filled out by the dentist. Their families (parents/guardians) will be asked to fill out the "Child Fear Assessment Scale-Dental Subscale (CFSS-DSc) before the session. 35 children will be included in the study. Main goal in this sesion is to evaluate in which dental practice step can be progressed in an anxious child by using classical behavior managament technique.

INTERVENTIONS:
Other: Pediatric Quiz Game — Investigator will start interacting with children upon their arrival and during their presence in the waiting room before entering the operating room. This will help to obtain better cooperation (frankl scale) and anxiety reductions (FIS and VPT) at different stages of the dental examination (e.g., entering the clinic, sitting on the dental chair, opening mouth, examination with mirror, probe, use of low-high-speed handpieces, ITR restoration). Pediatric Quiz is actually an ice-breaking quiz game developed for children, with the promise of a surprise gift at the end. It can be defined as "asking children basic questions on colors, animals, fruits and/or cities depending on the age of the child among which the child would choose him/herself and answer the question easily.
  Arms: Pediatric Quiz Game

SUMMARY:
Behavior orientation is the cornerstone of the success of pediatric dentistry. The use of behavior management techniques enables children to learn appropriate behavior and coping skills, reduce anxiety, and facilitate the delivery of adequate oral health care. Some behavior guidance systems have been tried to be created. On the basis of the magic game, it has been tried to move the children away from the current real situation, the reality of dental treatment, to move forward in communication and successful results have been obtained. The main thing in the technique is to start the communication with the child in the waiting room of the dentist and to reduce the anxiety of the child by improving the self-efficacy perception of the child. The aim of this study is to investigate the effectiveness of question-answer behavior guidance technique in dental treatment in pediatric patients.

DETAILED DESCRIPTION:
Behavior orientation is the cornerstone of the success of pediatric dentistry. The use of behavior management techniques enables children to learn appropriate behavior and coping skills, reduce anxiety, and facilitate the delivery of adequate oral health care. Better communication can be achieved when children feel the freedom to express themselves. In the same way, parents may state that in cases where there is no coercion and verbal communication, the children are uncomfortable and they have problems during their second-third dentist visits.

However, in some cases, success may not be achieved even if different behavior management techniques are applied. Activities such as diverting attention in children to other areas, starting the communication in the waiting room before entering the practice environment can lead to self-confidence, relaxation and confidence. The method of rewarding can also be very effective in directing behavior in children. For this reason, it communicates with a combination of some techniques without depending on only one technique and can lead to applications in dentistry practice.

Based on this idea, some behavior guidance systems have been tried to be created. On the basis of the magic game, it has been tried to move the children away from the current real situation, the reality of dental treatment, to move forward in communication and successful results have been obtained.

With this information, the aim of our study is to experience a new behavior management technique in children. The main thing in the technique is to start the communication with the child in the waiting room of the dentist and to reduce the anxiety of the child by improving the self-efficacy perception of the child. In this direction, in order to increase the child's self-efficacy perception, simple questions are asked to the child about colors, fruits and animals, if necessary, clues are given to give correct answers, and verbal praise for correct answers aims to increase self-efficacy perception and reduce anxiety. After the communication is started in the waiting room, the dental examination, dental chair and planned procedures will be introduced to the child, together with the tell-show-do method, as always practiced in the dental chair. The aim of this study is to investigate the effectiveness of question-answer behavior guidance technique in dental treatment in pediatric patients. Children's pain and anxiety levels were assessed by various tests designed to purpose. The Visual Analogue Scale (VAS), a self-reporting scale,was preferred to evaluate children's experience of pain. The scale displayed a colored spectrum on the front side ranging from no pain (white) to severe pain (red), which indicates relevant pain scores ranging from 0 to 10 on the reverse side.10

ELIGIBILITY:
Inclusion Criteria:

1. Children of age group 4-8 years.
2. with no previous dental experience.
3. without any systemic or mental disorders.

Exclusion Criteria:

1. Children or their families that could not agree to participate the study
2. They had a previous serious dental experience in need of emergency treatment
3. Having systemic or mental disorders

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | 3 Months
  Participants' pain and anxiety levels were assessed. The scale displayed a colored spectrum on the front side ranging from no pain (white) to severe pain (red), which indicates relevant pain scores ranging from 0 to 10 on the reverse side.
The Dental Subscale of Children's Fear Survey Schedule parental version (CFSS-DS pv) | 3 months
  The Scale consists of 15 articles. The answers are given by parents on a Likert type scale, ranging from 15 to 75. For children with moderate and severe dental fear levels, threshold values are set as 32 and 38 points, respectively.
The Venham Picture Test (VPT), a self-reporting scale | 3 months
  The scale is used to evaluate children's situational anxiety. It consists of 16 illustrations in pairs.Among the pairs, one represents the presence of anxiety and the other represents absence of anxiety. Children's anxiety scores were calculated between 0 and 8, according to the illustration they chose, representing themselves. Higher scores indicate the presence of anxiety and its level.
Facial Image Scale (FIS). | 3 months
  Self-report scale will be used in the study to evaluate children's state of anxiety. It displays nine faces showing emotions ranging from "non-anxious" to "very anxious." Participants are requested to indicate the face that represents their actual feelings. The scores range between 0.04 (positive/nonanxious) and 0.97 (negative/very anxious), demonstrating the state anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Faculty of Dentistry, Department of Pediatric Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shahnavaz S, Hedman-Lagerlof E, Hasselblad T, Reuterskiold L, Kaldo V, Dahllof G. Internet-Based Cognitive Behavioral Therapy for Children and Adolescents With Dental Anxiety: Open Trial. J Med Internet Res. 2018 Jan 22;20(1):e12. doi: 10.2196/jmir.7803. PMID 29358158
- [Result] Peretz B, Gluck G. Magic trick: a behavioural strategy for the management of strong-willed children. Int J Paediatr Dent. 2005 Nov;15(6):429-36. doi: 10.1111/j.1365-263X.2005.00668.x. PMID 16238653
- [Result] Grisolia BM, Dos Santos APP, Dhyppolito IM, Buchanan H, Hill K, Oliveira BH. Prevalence of dental anxiety in children and adolescents globally: A systematic review with meta-analyses. Int J Paediatr Dent. 2021 Mar;31(2):168-183. doi: 10.1111/ipd.12712. Epub 2020 Sep 9. PMID 33245591